CLINICAL TRIAL: NCT02867787
Title: Study of the Treatment of Tendinopathy Unruptured of Rotator Cuff by Intramuscular Injection of Botulinum Toxin
Acronym: Botox shoulder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Nicolas Pujol, Investigator coordinator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P13/09_ Botox
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Tendinopathy Rotator Cuff
Keywords: Shoulder Joint; A02.835.583.748

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botox arm (Experimental): intramuscular injection of botulinum toxin
  Interventions: Drug: Botox arm

INTERVENTIONS:
Drug: Botox arm

SUMMARY:
Botulinum toxin is used in musculoskeletal therapy routinely for 15 years. This is one of the most potent neurotoxins. It comes in 7 serotypes (A to G).Therapeutic application of botulinum toxin are mainly based on its ability to block the neuromuscular transmission by preventing the release of acetylcholine, creating paralysis muscle relative and reversible.

It has been used in the treatment of cervical dystonia, migraine headaches, and an antinociceptive effect. The analgesic effect occurred even prior to the release muscular. Several randomized studies have been published about it. The investigators assume that intramuscular injection of botulinum toxin is effective in the treatment of tendinopathy rotator cuff.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* Active social care
* Compliant patient with protocol
* Patient more than 18 years
* Positive Neer Test

Exclusion Criteria:

* Prior study exclusion period
* Protected patient
* Study refusal
* Deficient patient
* Rheumatoid arthritis, osteoarthritis, chondrocalcinosis.
* Microcrystalline arthritis.
* Active infection .
* History of hypersensitivity reaction during a previous injection of botulinum toxin
* Bilateral involvement
* Neurological deficit
* Depression
* History of shoulder surgery
* Pregnant or breast feeding women
* Systemic disease (diabeta, vascularitis)
* Known neurological disease
* Intraarticular associate disease
* Acromioclavicular associate disease
* Myasthenia
* Botulinum toxin is not recommended in combination with aminoglycosides

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Significant improvement in shoulder pain objectified by analogy Visual Scale (VAS) in patients with unruptured tendinopathy of the rotator cuff impingement, debilitating, lasting for more than 3 months and resistant to usual medical treatment. | 3 months

SECONDARY OUTCOMES:
Significant improvement in life quality : functional clinical scores (Constant, ASES, Oxford) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pujol Nicolas, MD, Principal Investigator — CH Versailles
Locations (1):
- CH Versailles, Le Chesnay, France